CLINICAL TRIAL: NCT06821802
Title: Effect of Protein Supplementation in Hospitalized Patients With Hyponatremia Due to the Syndrome of Inappropriate Antidiuresis - a Monocentric Randomized Open-label Pragmatic Active-controlled Trial - the TREASUREx Trial
Brief Title: Protein Supplementation in Hyponatremia Due to the Syndrome of Inappropriate Antidiuresis
Acronym: TREASUREx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-02282; kt25ChristCrain2
Record Dates: First submitted 2025-01-30; First posted 2025-02-12 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Hyponatremia; Syndrome of Inappropriate Antidiuresis
Keywords: dysregulated arginine vasopressin (AVP) secretion; increased renal AVP sensitivity; protein supplementation; fluid restriction
MeSH Terms: conditions — Hyponatremia; Inappropriate ADH Syndrome; Diabetes Insipidus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein Supplementation (Experimental): 80 g protein supplementation per day (two bottles, each containing 40 g protein)
  Interventions: Dietary Supplement: Moltein PURE Protein Powder
- Fluid restriction (Active Comparator): total daily fluid intake to a maximum of 1000 ml
  Interventions: Behavioral: Fluid restriction

INTERVENTIONS:
Dietary Supplement: Moltein PURE Protein Powder — 80 g protein supplementation per day (two bottles, each containing 40 g protein)
  Arms: Protein Supplementation
Behavioral: Fluid restriction — total daily fluid intake to a maximum of 1000 ml
  Arms: Fluid restriction

SUMMARY:
The goal of this study is to assess the impact of protein supplementation on hyponatremia caused by the syndrome of inappropriate antidiuresis during hospitalization.

DETAILED DESCRIPTION:
Hyponatremia (plasma sodium <135 mmol/L) is the most common electrolyte disorder, affecting up to 30% of hospitalized patients. Chronic hyponatremia (>48 hours) is linked to longer hospital stays, higher costs, increased mortality, and morbidity (e.g., falls, fractures, cognitive deficits). The most common cause of euvolemic hyponatremia is syndrome of inappropriate antidiuresis (SIAD), characterized by excessive water retention due to dysregulated vasopressin activity. Treatment options include fluid restriction or increasing water excretion with AVP antagonists, SGLT2 inhibitors, or oral urea.

A recent trial showed that protein supplementation can induce osmotic diuresis and raise sodium levels similarly to oral urea, with better tolerability. Since protein supplementation is often used in hospitalized patients with malnutrition, this study aims to compare its acceptability to fluid restriction in hospitalized SIAD patients. This head-to-head superiority trial will randomize patients to receive either 80 g of dietary protein daily or fluid restriction (1000 mL/day) for up to 5 days. The hypothesis is that protein supplementation is significantly more acceptable to patients than fluid restriction, ultimately improving treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with confirmed SIAD during the hospital stay or at screening, defined by:
* Plasma sodium concentration <135 mmol/L
* Plasma osmolality <300 mOsm/kg
* Urine osmolality >100 mOsm/kg
* Urine sodium concentration >30 mmol/L
* Clinical euvolemia (no signs of hypovolemia or hypervolemia)

Exclusion Criteria:

* Lactose intolerance, milk protein allergy, soy allergy, nuts allergy, or hypersensitivity to components of the protein supplement.
* Inborn metabolic disorders affecting carbohydrate, lipid, or protein metabolism.
* Severe symptomatic hyponatremia requiring 3% NaCl or intensive care.
* New (within the last five days) treatment with SGLT2 inhibitors, vaptans or oral urea
* Uncontrolled severe hypothyroidism (untreated)
* Uncontrolled adrenal insufficiency (morning cortisol <150nmol/l)
* eGFR <45 mL/min/1.73 m² (KDIGO G3b-5) or end-stage renal disease (dialysis)
* Severe hepatic impairment or advanced symptomatic liver disease defined as past or current hepatic encephalopathy, liver cirrhosis Child C, or decompensated (bleeding, jaundice, hepatorenal syndrome)
* Pregnancy, breastfeeding, or plans to become pregnant during the study.
* End-of-life care
* Lack of capacity or other reasons preventing from giving informed consent or following study procedures (e.g., due to language problems, psychological disorders, dementia, etc.)
* Treatment with thiazid diuretic (must be stopped at least 48 hours before inclusion)

Post-randomization Exclusion Criteria:

* Type 1 diabetes or uncontrolled type 2 diabetes (HbA1c >8.0%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure (AIM) questionnaire | On day 5 (or discharge)
  Treatment acceptability is assessed using the Acceptability of Intervention Measure (AIM) questionnaire, a validated patient-reported outcome measure scored on a 1 to 5 Likert scale. The total AIM score ranges from 4 to 20, with higher scores indicating greater acceptability. The primary analysis will compare AIM scores between the two treatment groups at the end of the intervention (day 5 or discharge).

SECONDARY OUTCOMES:
Plasma sodium levels | Daily measurements from the day of inclusion to day 5
  Change in change in plasma sodium levels in mmol/l will be assessed at study inclusion to day 5 of treatment or until discharge
Estimated glomerular filtration rate (eGFR) | On the day of inclusion and on day 5
  Assessement of creatinine levels
Changes in blood electrolytes | On the day of inclusion and on day 5
  Assessement of sodium levels
Changes in urine electrolytes | On the day of inclusion and on day 5
  Assessement of sodium levels
Changes in glucose levels | On the day of inclusion and on day 5
  Assessement of glucose levels
Changes kidney parameters | On the day of inclusion and on day 5
  Assessement of urea and uric acid levels
Plasma sodium levels one day after treatment start | On the day of inclusion and 12-36 hours after treatment initiation
  Plasma sodium levels 12-36 hours after treatment start in patients with a plasma sodium concentration <125 mmol/L at baseline.
Endocrine parameters | On the day of inclusion and on day 5
  Blood levels of copeptin, aldosterone, renin, MR-proANP and NT-proBNP, apelin, etc. are assessed
General well-being | On the day of inclusion and on day 5
  General well-being measured by numerical rating scale (NRS). Score from 0-10 while 10 indicates improved well-being
Symptoms of hyponatremia | On the day of inclusion and on day 5
  Symptoms of hyponatremia (e.g. vertigo, headache, nausea, attention deficit, mental slowness, forgetfulness, gait instability) assessed by a questionnaire (yes/no; if yes: VAS, 0-10).
Fluid intake | Daily measurements from the day of inclusion to day 5
  Oral daily fluid intake assessed using a self-completed drinking protocol.
Changes in body weight | On the day of inclusion and on day 5
  Body weight is assessed
Changes in blood pressure | On the day of inclusion and on day 5
  Systolic and diastolic blood pressure will be measured
Changes in heart rate | On the day of inclusion and on day 5
  Heart rate will be assessed
Differences in clinical outcomes - length of hospital stays | Daily from the day of inclusion to day 5
  Length of hospital stays will be assessed
Need for additional hyponatremia treatment and treatment escalation | Daily from the day of inclusion to day 5
  Assessment of treatment escalation (YES/NO) including: A: administration of 3% NaCl infusion; B: administration of oral urea; C administration of SGLT2 inhibitors; D: administration of vaptans; E: administration of diuretics; F: other during the treatment period.
Treatment compliance | Daily from the day of inclusion to day 5
  The participant's daily consumption of protein drinks and/or their adherence to a fluid restriction regimen is recorded.
Quality of life (EQ-5D-5L) questionnaire | On the day of inclusion and on day 5
  Participants' health-related quality of life is assessed using the EuroQol 5 Dimensions, 5 Levels (EQ-5D-5L) questionnaire. , which includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on five levels, ranging from no problems to extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof. MD, Principal Investigator — Universitätsspital Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland